CLINICAL TRIAL: NCT02245178
Title: Lung Function Decline and Disease Risk From Young Adulthood to Middle Age
Acronym: CARDIA Lung
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Minnesota (Other); University of Alabama at Birmingham (Other); University of Kentucky (Other); Kaiser Foundation Research Institute (Other); Brigham and Women's Hospital (Other); Vanderbilt University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ravi Kalhan, Associate Professor, Northwestern University
Other Study IDs: STU00090966; R01HL122477 (NIH)
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: COPD; Lung Function; Heart - Lung Interaction; Restrictive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obervational - CARDIA participants: CARDIA study participants will undergo lung function testing and have existing thoracic CT scans analyzed for lung structure.
  Interventions: Procedure: Lung spirometry; Other: CT scan analysis

INTERVENTIONS:
Procedure: Lung spirometry — measurement of pulmonary function pre- and post-bronchodilator
  Other Names: lung function
Other: CT scan analysis — Analysis of existing year 25 thoracic CT scans for lung and intrathoracic vascular structure

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death in the United States, but markers that predict risk of developing disease outside of cigarette smoking have not been identified. Individuals with lung disease frequently have concurrent cardiovascular disease, but the reason for this is not well understood. In this study, we will identify markers that predict risk of future lung disease and evaluate the concurrent subclinical evolution of lung and heart dysfunction. This will allow for targeting of preventive strategies to stop the rising incidence of COPD and other lung diseases and provide insights into why heart and lung disease frequently occur together.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death in the United States. Although smoking is a major risk factor for COPD, only a minority of smokers develops COPD. Markers that predict risk of future COPD in young adults would be valuable to target risk reduction strategies and identify subclinical disease. Although COPD is classically defined by obstructive lung physiology, many individuals, including smokers, have spirometric restrictive physiology. Reduced lung function, whether manifesting as COPD or restriction, is associated with adverse cardiovascular outcomes. Our long-term goals are to identify subclinical manifestations of COPD and other lung disease and explore why heart and lung disease co-exist. This is an ancillary study to the Coronary Artery Risk Development in Young Adults (CARDIA) cohort study's year 30 examination. We will add pre- and post-bronchodilator spirometry to the exam and evaluate the lung parenchymal and vascular structure on cardiac CT scans from year 25. Informed by our preliminary data which documents that markers of systemic inflammation and endothelial dysfunction are associated with subsequent lung function decline in young adults, that lung function decline in young adults is associated with incident hypertension, and that there is a divergence in cardiac structure and function depending on the pattern of lung function decline, we propose the following specific aims: (1) To evaluate factors in young adults that predict incident COPD and/or restriction; (2) To determine whether incident COPD and incident restriction are associated with distinct cardiac structural and functional changes; and (3) To determine the lung structural and intrathoracic vascular changes associated with incident COPD and incident restriction. We will test the hypothesis that early life markers of systemic inflammation and endothelial dysfunction are associated with risk of subsequent lung disease and explore whether different inflammatory markers predict different lung phenotypes. We will then evaluate the cardiac structural changes associated with different lung phenotypes and evaluate the lung structural and pulmonary vascular alterations that may explain the concurrently evolving cardiovascular findings associated with developing lung disease. These studies will describe the subclinical manifestations of lung disease, identify markers that predict risk of future lung disease, and expand our understanding of heart-lung interactions as they evolve from health in young adults to disease in middle age.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the main CARDIA examination at year 30

Exclusion Criteria:

* Shortness of breath with pain in the chest within the past week
* Heart attack or stroke within the past month

Ages: 48 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in the main Coronary Artery Risk Development in Young Adults (CARDIA) cohort study attending the year 30 examination
Sampling Method: Non-Probability Sample
Enrollment: 3193 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Incident COPD | 30 years
  From cohort initiation, predictors of incident COPD

SECONDARY OUTCOMES:
Incident restriction | 30 years
  From cohort initiation, predictors of incident restrictive lung physiology

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kalhan, MD, Principal Investigator — Northwestern University